CLINICAL TRIAL: NCT04857957
Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CNTX-6016 in Healthy Subjects and a Single Cohort of Subjects With Painful Diabetic Neuropathy
Brief Title: Safety, Tolerability & Pharmacokinetics Study of CNTX-6016 in Healthy Subjects and Subjects With PDN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNTX-6016o-HV/PDN-102
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2023-10

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): Dose 1
  Interventions: Drug: Oral dose CNTX-6016 or oral dose Placebo
- Cohort 2 (Experimental): Dose 2
  Interventions: Drug: Oral dose CNTX-6016 or oral dose Placebo
- Cohort 3 (Experimental): Dose 3
  Interventions: Drug: Oral dose CNTX-6016 or oral dose Placebo
- PDN cohort (Experimental): Dose based on safety in healthy Cohorts 1-3
  Interventions: Drug: Oral dose CNTX-6016 or oral dose Placebo

INTERVENTIONS:
Drug: Oral dose CNTX-6016 or oral dose Placebo — CNTX-6016 or Placebo

SUMMARY:
A Phase 1b study to evaluate the safety, tolerability and pharmacokinetics of multiple ascending doses of CNTX-6016 in healthy subjects and a single cohort to evaluate painful diabetic neuropathy.

ELIGIBILITY:
Key Inclusion Criteria:

* Is in good general health as determined by Investigator's review.
* Has a body mass index (BMI) between 18 and 35 kg/m2.
* Non- or ex-smoker (> 1 year) and has not used any nicotine containing products within 12 months prior to screening.
* For females, is not currently pregnant and is either of non-childbearing potential or willing to use an adequate method of birth control.
* For males, must agree to use barrier contraception and not to donate sperm

Key Exclusion Criteria:

* Is pregnant, lactating, or planning a pregnancy during the study.
* Tests positive for COVID-19 after screening is complete and subject is confirmed to enroll
* History of or active cardiac disease, including congestive heart failure, angina, or any arrhythmia.
* Has any history or currently active type of cancer except excised or cured basal cell carcinoma.
* Has an immunological disorder such as, but not limited to, human immunodeficiency virus (HIV), acquired, or congenital immune deficiency syndrome; autoimmune diseases, such as, but not limited to, rheumatoid arthritis, systemic lupus erythematosus, seronegative spondyloarthropathies or vasculitis, or any infection.
* Positive urine screen for alcohol, cotinine, THC and/or drugs of abuse
* Has positive screening test for hepatitis B virus (HBV) or hepatitis C virus (HCV).

Key Inclusion Criteria- PDN Cohort

* A diagnosis/history of Type 2 diabetes mellitus
* The pain is present in both feet/legs with symmetrical onset
* The pain is characterized as burning, painful, cold or electrical shocks in nature
* The pain is associated with tingling, numbness, itching or pins and needles type sensations
* The pain has been present and consistent for ≥ 6 months

Key Exclusion Criteria- PDN Cohort

* Diagnosis of Type 1 diabetes
* Has serious or unstable cardiovascular, hepatic, renal, respiratory or hematological illness
* Has a history or currently active type of cancer except excised or cured basal cell carcinoma.
* Has a History of psychological conditions or neurological disorders
* Has a History of lower back pain with radiculopathy
* Has received non-pharmacological treatment for pain within 14 days
* Has a history of frequent and/or severe allergic reactions with multiple medications

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) (safety and tolerability) with CNTX-6016 | Up to 45 days
  Number of participants with TEAEs, which includes laboratory test variables
CNTX-6016 Pharmacokinetics - Cmax | Up to Day 6
  Systemic exposure to CNTX-6016 measured by Cmax
CNTX-6016 Pharmacokinetics - AUC0-t | Up to Day 6
  Systemic exposure to CNTX-6016 measured by AUC0-t
CNTX-6016 Pharmacokinetics - t1/2 | Up to Day 6
  Systemic exposure to CNTX-6016 measured by t1/2
CNTX-6016 Pharmacokinetics - tmax | Up to Day 6
  Systemic exposure to CNTX-6016 measured by tmax

OTHER OUTCOMES:
CNTX-6016 Effect of Age and Sex in all Cohorts | Up to Day 14
  Systemic exposure to CNTX-6016 By Cmax pooled from all cohorts over full dose range.
CNTX-6016 Effect of Age and Sex in all Cohorts | Up to Day 14
  Systemic exposure to CNTX-6016 By AUC pooled from all cohorts over full dose range.
CNTX-6016 Efficacy - PDN Cohort | Up to Day 14
  Efficacy measured by Numeric Rating Scale. The Numeric Rating Scale is an 11-point pain scale with a range of 0 to 10 where 0 = "no pain" and 10 = "worst possible pain"
CNTX-6016 Efficacy - PDN Cohort | Up to Day 14
  Efficacy measured by PainDETECT Questionnaire
CNTX-6016 Efficacy - PDN Cohort | Up to Day 14
  Efficacy measured by Patient Global Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Randall Stevens, MD, Study Chair — Centrexion Therapeutics
Locations (1):
- AltaSciences, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No